CLINICAL TRIAL: NCT04809753
Title: Eustachian Tube Dilation Using an Angioplasty Balloon - a Pilot Safety Study
Brief Title: Eustachian Tube Dilation With an Endovascular Balloon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3776
Record Dates: First submitted 2021-02-24; First posted 2021-03-22 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Eustachian Tube Dysfunction; Eustachian Tube Dysfunction of Both Ears

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eustachian tube dilation (Experimental): Eustachian tube dilation with an endovascular balloon
  Interventions: Device: Eustachian tube dilation

INTERVENTIONS:
Device: Eustachian tube dilation — Dilation of the eustachian tube with an endovascular balloon

SUMMARY:
The Eustachian tube is a narrow tube which links the back of the nose to the middle ear. Eustachian tube dysfunction may occur when the mucosal lining of the tube is swollen, or does not open or close properly. It can occur after the start of a cold and other nose, sinus, ear and throat infections causing ear pain and pressure, fullness, cracking/popping sounds. This is an ubiquitous healthcare problem, affecting children and adults, that can lead to severe consequences including hearing loss, chronic otitis media, tinnitus, and vertigo. Numerous studies have consistently failed to support the effectiveness of medical managements. Pressure equalizing tubes are considered a temporary solution that does not treat the underlying pathology. More recent preliminary evidence of using inflation of a noncompressible balloon in the eustachian tube improved clinical outcomes, patients' symptoms and quality of life. This eustachian dilation catheter is not accessible in Canada since the device and procedure is not covered by OHIP (Ontario health insurance plan) or any other health insurance in Canada. In a cadaver study, we have evaluated using an endovascular balloon (Balloon that is used to dilate (expand) vessels) for eustachian tube dilation, which only costs about 10% of the eustachian tube dilation device. This endovascular balloon is Health Canada approved, but not for this specific use. We therefore want to conduct a pilot safety study with the main goal of assessing feasibility of eustachian tube dilation with the endovascular device.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old (of both sexes)
* Diagnosed with unilateral or bilateral persistent obstructive eustachian tube dysfunction (OETD)
* Undergoing tympanoplasty or tympanomastoidectomy

Exclusion Criteria:

* Patulous eustachian tube
* Preoperative nasal endoscopy with evidence of anatomic conditions that would prevent transnasal access to the Eustachian tube
* CT temporal bone scan with evidence of carotid artery dehiscence, superior semicircular canal dehiscence, or extrinsic eustachian tube compression
* Patient unable to follow protocol for any reason
* Cleft palate or Craniofacial syndrome
* Prior eustachian tube intervention
* Prior radiation to the head and neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Succesfull procedure | 20 minutes
  o Feasibility to perform the procedure after ear surgery with no local complication and within 15-20 minutes

SECONDARY OUTCOMES:
CT | 5 minutes
  o Safety evaluated after the procedure CT scan. Complications (adverse and serious adverse events related to the device or procedure)
ETDQ - 7 (Eustachian Tube Dysfunction Questionnaire - Item 7) | 2 minutes
  o Mean change in overall ETDQ-7 scores from baseline at 2- and 6-months follow-up
Endoscopic evaluation | 5 minutes
  Safety evaluated after the procedure by endoscopic examination and CT scan. Complications (adverse and serious adverse events related to the device or procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Trung Le, MD, Principal Investigator — Sunnybrook Health Sciences Center
Locations (1):
- Sunnybrook Health Sciences Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data (consent form (anonymized), study protocol) will be shared upon reasonable request after publication

REFERENCES:
- [Derived] Dahm V, Lui JT, Jung S, Lin VY, Chen JM, Le TN. The feasibility and safety of eustachian tube dilation with a standard endovascular balloon: a clinical pilot study. J Otolaryngol Head Neck Surg. 2023 Feb 28;52(1):20. doi: 10.1186/s40463-022-00599-1. PMID 36855202